CLINICAL TRIAL: NCT06723223
Title: Clinical Validation of a Combined Equilibration Test in Patients on Peritoneal Dialysis
Brief Title: Novel Combined Function Test for Patients on Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CPET202002377
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: End Stage Kidney Disease (ESRD)
Keywords: Peritoneal dialysis; Peritoneal equilibration test; CombiPET
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients (Experimental)
  Interventions: Diagnostic Test: Traditional Peritoneal Equilibrium Test; Diagnostic Test: Combined Peritoneal Equilibrium Test

INTERVENTIONS:
Diagnostic Test: Traditional Peritoneal Equilibrium Test — The first day started with a traditional PET consisting of a 240-minutes dwell with 2.3% glucose PD solutions. The intervention includes sampling of blood plasma (Na, K, glucose, creatinine, urea and albumin) and dialysate (Na, K, glucose, creatinine, urea and albumin).
Diagnostic Test: Combined Peritoneal Equilibrium Test — The PET test on the first day (Day 1) was followed by a short (60 min) combined PET with 4.25% glucose solution. On the second day (Day 2), the combined PET was repeated. The intervention includes sampling of blood plasma (Na, K, glucose, creatinine, urea and albumin) and dialysate (Na, K, glucose, creatinine, urea and albumin).

SUMMARY:
Peritoneal membrane function tests such as the traditional peritoneal equilibrium test (PET) aid in the assessment of various peritoneal membrane functions, and are widely used in clinical practice to guide dialysis prescription, and also to monitor the integrity of the peritoneal membrane over time. Traditional tests do however have several shortcomings such as being time consuming, complex, and having a low reliability. Also, present functional tests often provide limited information such as small solute transfer rates, which means that other functional changes go unnoticed.

The present study investigates the reliability of a novel short (60 min) test, with the potential of replacing complex and time-consuming conventional tests. The novel test provides a comprehensive assessment on both water- and solute transfer across the peritoneal membrane, including the osmotic conductance to glucose (OCG), small solute diffusive conductance (in terms of the diffusive surface to diffusion length ratio, A0/Δx), and also macromolecular transport and apparent fluid absorption. In contrast to conventional tests, multiple fill volumes may be used and results are also applicable to all glucose strengths used in conventional peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis treatment duration of at least 1 month
* No recent peritonitis (a minimum of 1 month since the last peritonitis)

Exclusion Criteria:

* Pregnancy
* Participant unable to provide informed consent
* Peritonitis
* Other acute infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Reliability of the combined peritoneal equilibrium test | All interventions need to be completed within one month.
  Reliability of the novel test will be assessed using the Intraclass Correlation Coefficient (ICC) evaluating consistency and repeatability of key continuous measurements (osmotic conductance to glucose, diffusive conductance, albumin clearance, and apparent fluid absorption) across the two different test occasions (Day 1 and Day 2)

SECONDARY OUTCOMES:
Comparison of the Traditional vs. Combined Peritoneal Equilibrium Test | All interventions are performed within one month.
  The key continuous outcome measures (osmotic conductance to glucose and diffusive conductance) from the combined peritoneal equilibrium test (PET) will be inserted into the isocratic model (and the three-pore model) for peritoneal dialysis to test if the results in the traditional PET can be accurately reproduced. The rationale is to elucidate if the combined PET contains the same information as the tradional PET or if information is lost in the much shorter combined PET.

CONTACTS AND LOCATIONS:
Overall Officials: Carl M Öberg, M.D., Ph.D., Principal Investigator — Lund University
Locations (1):
- Hemdialysmottagningen, Skånes Universitetssjukhus (SUS) Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided